CLINICAL TRIAL: NCT03086785
Title: Prospective, Multicenter, Observational Study of Apatinib Single or Combined Capecitabine for Treatment of Patients With Metastatic Her-2 Negative Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hebei Medical University Fourth Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HB-B001
Record Dates: First submitted 2017-03-16; First posted 2017-03-22 (Actual); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Breast Cancer Metastatic
MeSH Terms: interventions — apatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- apatinib (Experimental): apatinib 500mg qd po or combined Capecitabine 1000mg/m2 bid d1-d14 q3w
  Interventions: Drug: Apatinib

INTERVENTIONS:
Drug: Apatinib — apatinib 500mg qd po or combined capecitabine 1000mg/m2 bid d1-14 q3w

SUMMARY:
The purpose of this study is to assess the efficacy and safety of patients who receive apatinib single or combined capecitabine for treatment of patients with metastatic her-2 negative breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 70 years old (female)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Pathologically diagnosed with her-2 negative, ER/PR negative, ER/PR positive after the failure of endocrine treatment, and had not more than three chemotherapy regimens (must include anthracycline-based and yew class), and the final failure of chemotherapy regimens in patients with advanced breast cancer; Note: treatment failure include (1) during or after the completion of six months or less disease progress of neoadjuvant or adjuvant therapy; (2) rescue treatment in progress within 3 months or less
* Patients with at least one measurable lesions of the advanced breast cancer， measurable lesions has not received radiotherapy or other treatment, unless progress after treatment (measuring≥10mm on spiral CT scan, satisfying the criteria in RECIST1.1 and WHO);
* Major organ function has to meet the following certeria:

  1. For results of blood routine test (without blood transfusion within 14 days)

     1. HB≥100g/L;
     2. ANC≥1.5×109/L;
     3. PLT≥75×109/L;
  2. For results of blood biochemical test：

     1. TBIL<1.5ULN；
     2. ALTand AST<2.5ULN, but5<ULN if the transferanse elevation is due to liver metastases；
     3. Serum creatinine ≤1.25ULN , or calculated creatinine clearance>45 ml/min(per the Cockcroft-Gault formula); 6.Participants were willing to join in this study, and written informed consent.

Exclusion Criteria:

1. The patients with the failure of capecitabine treatment；
2. The patients with chest wall invasion, or chest wall large canker has a tendency to transfer；
3. Have high blood pressure and antihypertensive drug treatment can not control (systolic blood pressure > 140 mmHg, diastolic blood pressure > 90 mmHg), with classⅡand above coronary heart disease, unable to control arrhythmia (including QTc lengthened women > 470 ms) and classⅢ-Ⅳcardiac insufficiency; or Left ventricular ejection fraction (LVEF) < 50%；
4. A variety of factors influencing oral drugs (such as unable to swallow, after resection of the gastrointestinal, chronic diarrhea and intestinal obstruction, etc.)；
5. Has a history of bleeding, the clinical significance of bleeding symptoms, patients with definite bleeding tendency, such as gastrointestinal bleeding, bleeding ulcers, baseline period （+ +）and above of defecate occult blood, vasculitis, etc；
6. Received a major surgery within 4 weeks or severe traumatic injury, fractures, or has a poor healing wound；
7. Allergic to apatinib and supplementary material；
8. Patients with active brain metastases;
9. Patients with pregnant or planning a pregnancy;
10. The researchers think inappropriate.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-11-24 (Actual); Primary Completion 2018-11 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | evaluated in 24 months since the treatment began
  Baseline to measured date of progression or death from any cause

SECONDARY OUTCOMES:
Overall survival | the first day of treatment to death or last survival confirm date,up to 24 months
  Baseline to measured date of death from any cause
Disease control rate | tumor assessment every 6 weeks since the treatment began，up to 24 months
  Baseline to measured progressive disease
Objective response rate | tumor assessment every 6 weeks since the treatment began，up to 24 months
  Baseline to measured stable disease
Side effects | evaluated in the 24th month since the treatment began according to the Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0
  throughout study

CONTACTS AND LOCATIONS:
Overall Officials: cuizhi Geng, archiat, Principal Investigator — Hebei Medical University Fourth Hospital; zefei Jiang, archiat, Principal Investigator — The 307th Hospital of Chinese Peoples' Liberation Army
Locations (1):
- Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei, China